CLINICAL TRIAL: NCT04044456
Title: Combining Attention and Metacognitive Training to Improve Goal Directed Behavior in Veterans With TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N3189-P
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Brain Injury; Cognition; Veteran; Attention; Metacognition
MeSH Terms: conditions — Brain Concussion; Brain Injuries | interventions — Motion Pictures

STUDY DESIGN:
Intervention Model Description: participants meeting inclusion criteria will be randomized to either treatment (Goal management training and attention training) or control (Brain Health Workshop and national geographic movies).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GMT plus attention (Experimental): GMT consists of 2-hour, 10 weekly sessions using an interactive Power Point presentations. Attention training consists of 2-hour computerized attention training using Attention Process Training III and Brain HQ.
  Interventions: Behavioral: Goal Management Training; Behavioral: Attention Training
- BHW plus movies (Placebo Comparator): Brain Health Workshop consists of 2-hour, 10 weekly sessions using Power Point presentations and national geographic movies (2-hour, 10 weekly sessions).
  Interventions: Behavioral: Brain Health Workshop; Behavioral: National geographic movies

INTERVENTIONS:
Behavioral: Goal Management Training — GMT: is a 10-session intervention to improve planning and problem solving. Interactive Power Point modules are administered by a cognitive therapist. Each session builds on the steps of a five-stage planning and problem-solving strategy. Veterans will be taught to generate and verbalize the following five-steps: "stop-what am I doing?", "define the goal", "list the steps", "learn the steps"; then, "check-am I doing what I planned?" The five-stage strategy is then incorporated into a variety of activities in the laboratory and in-home assignments.
  Other Names: GMT
  Arms: GMT plus attention
Behavioral: Attention Training — Attention Process Training (APT-III) will be administered for a second weekly session in addition to the GMT session. Each session will be 2 hours/ week for 10 weeks. Veterans will also engage in BrainHQTM attention training at home for one-hour, five days/ week comprised of selected components of BrainHQ from Posit Science Corporation. This web-based computerized CRT modality of cognitive training is a restorative or "bottom-up" approach that targets basic cognitive skills such as arousal and vigilance processes, attention and information processing, and directly engages fundamental attention-control skills through repetitive graded exercises.
  Other Names: APT III, Brain HQ
  Arms: GMT plus attention
Behavioral: Brain Health Workshop — . BHW was developed specifically for consistency with GMT session length and contact with the facilitator49. BHW is an education presentation on brain function and cognitive principles of learning with homework and quizzes on information covered. To match time and contact of attention training, control participants will meet with the therapist for a separate two-hour session from BHW
  Other Names: BHW
  Arms: BHW plus movies
Behavioral: National geographic movies — participants will select movies to watch and answer a few questions about to equate the time and therapist interaction to attention training in arm 1.
  Other Names: movies
  Arms: BHW plus movies

SUMMARY:
Veterans with mild traumatic brain injury continue to deal with symptoms that interfere with their ability to engage in productive activities. In combination with other psychosocial difficulties, impairments are found in cognition, such as attention and executive function. Few interventions are available to treat attention in Veterans with mTBI. Of the interventions available, none rigorously train attention combined with strategy training. This project will innovatively combine a strategy training called Goal Management Training with computerized attention training to improve tests of problem solving, attention and functional tasks compared to a control group.

DETAILED DESCRIPTION:
This is a pilot study to test the effect of GMT plus Attention Training for Veterans with chronic mTBI. The research design is a parallel study with randomization to treatment or control with test administration at pre/post and six months following treatment. The investigators will enroll 50 Veterans with a diagnosis mTBI between the ages of 18 to 55, that demonstrate a deficit in attention, pass effort testing and have not changed psychotropic medication within the past two weeks. Treatment utilizes GMT for 10-weekly two-hour sessions and Brain HQ/Attention Process Training III for 10-weekly two-hour sessions. Control utilizes a complimentary Brain Health Workshop for 10-weely two-hour sessions and National Geographic movies for 10-weekly two-hour sessions.

Aim 1: Determine the treatment effect of attention training combined with GMT in Veterans with mTBI.

Hypothesis 1: GMT plus attention training will significantly improve performance on tests of cognition compared to the control group.

Primary measure: Computerized Tower of London (cTOL) total time, time to first move and optimal moves). The investigators have found significant improvement in cTOL following GMT in previous cohorts of Veterans with blast-related mTBI and anticipate improvement following a combined intervention.

Secondary measure: Attention Network Task (ANT) reaction time and errors for one or all dissociable components of three attentional systems (orienting, alerting, executive control) following intervention. There is little understanding of components of impaired attention and how it impacts executive function; therefore, there is limited guidance in shaping cognitive training. The investigators will conduct an experimental task (attention network task) that disassociates three attentional components (alerting, orienting, and executive control). The investigators will specifically target the orienting component of attention that is problematic for Veterans with mTBI and PTSD24, 26. Attentional processes are vital to goal-directed behavior. There is great potential in the use of these measures to identify individual differences (type of attention deficit) that could moderate treatment-related improvement and inform targeted interventions.

Hypothesis 2: Treatment gains will translate to functional activities compared to controls.

Primary measure of functional performance: test of grocery shopping skills (TOGSS) total time and optimal strategy use. The TOGSS captures efficiency in completing a real-world task and aligns with the strategy skills learned in GMT.

Secondary measure of community participation, the Community Reintegration of Servicemembers (CRIS) extent of participation. The CRIS demonstrated significant GMT treatment effect compared to controls in Veterans with mTBI. The combined treatment of attention training using drill training and implementing strategies to improve attention in a functional setting through GMT will potentiate treatment effect to functional activities. Measuring functional improvement through performance-based measures and self-report of engagement in activities will demonstrate treatment translation.

Tertiary analysis will be conducted on moderator variables: PTSD symptoms, Pain, History of Substance Abuse, Depression, number of concussions and combat exposure.

Successful completion of the proposed study will provide insight into the effectiveness of the innovative combined treatment of attention and executive function in Veterans with mTBI and PTSD. Use of the ANT could better target treatment and lead to future examination of attention treatment on neuroplasticity.

A multiple linear regression model will be used to determine if there is a significant association between treatment effect and comorbidities such as PTSD, depression, anxiety, pain, sleep, substance abuse, etc.

ELIGIBILITY:
Inclusion Criteria:

Veterans with a diagnosis mTBI between the ages of 18 to 55, that demonstrate a deficit in attention, pass effort testing and have not changed psychotropic medication within the past two weeks.

* all Veterans who have served in OIF-OEF-OND with single- (at least brief loss of conscious) or multiple (with at least alteration of consciousness) mild traumatic brain injury (mTBI) during deployment, who seek services at North Florida/South Georgia Veterans Health System (NF-VHS).
* TBI must have suffered their injury at least 6 months prior to study enrollment and currently be in stable neurological condition.
* age range 19-55 years to reduce the impact of aging on treatment improvement.
* Attention deficit of 1.5 SD below the mean of the RBANS attention index. This will ensure that participants have an objective deficit attention.
* Family member or friend that is willing to complete the BRIEF-A (BRIEF-A guidelines of face to face interaction with the participant at least twice a week) at all measurement time points.
* Access to a home computer, or smartphone with internet access.

Exclusion Criteria:

* History of pre-morbid learning disability
* History of psychiatric diagnosis sufficiently severe to have resulted in inpatient hospitalization.
* Neurological disease unrelated to TBI (seizure disorder, stroke)
* Score < 90 on National Adult Reading Test (NART)
* Failure of validity testing on either the Test of Memory Malingering (TOMM),). Score of 45 or less on TOMM Trial 2 or retention trial.
* Reported alcohol or substance abuse within the past year
* Reported involvement in current litigation
* Recent change of medications for seizures, depression or memory.
* Currently enrolled in other cognitive therapy that cannot be discontinued
* Does not speak English fluently
* Not competent to provide consent (also, not able to demonstrate understanding of expectations of study and potential risks of participation).
* Uncontrolled, acute medical or psychiatric condition as indicated by the participant or observed by the research team member that would make it unsafe to participate in the research activities, i.e. precautions for active homicidal/suicidal intent, active psychosis, or acute symptoms requiring immediate medical attention.
* Psychotropic drugs that have changed within the past two-weeks that would impact performance during assessment.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia K. Waid-Ebbs, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GMT Plus Attention | BHW Plus Movies
Started | 18 | 2
Completed | 13 | 1
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Veterans with mild traumatic brain injury
Groups:
- Total: Total of all reporting groups
Arm/Group | GMT Plus Attention | BHW Plus Movies | Total
Number analyzed (Participants) | 18 | 2 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: number analyzed were participants that completed treatment
  years
    number analyzed (Participants) | 13 | 1 | 14
    (all) | 42 (6.54) | 38 (0) | 42 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 15 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 17 | 1 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 1 | 11
  White | 8 | 1 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Computerized Tower of London Average Time to Complete Problems/Total Time
Description: Computerized Tower of London (cTOL) total time, week 1, week 11 and week 36. Complete game board of three colored balls to match goal board in the least amount of moves and as quickly as possible. range of total time is 0-59 seconds with lower time=better performance.
Time Frame: week 1, 11, 36
Population: Veterans with mild TBI that completed GMT training and 1 Veteran with mild TBI that completed the control sessions.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | GMT Plus Attention | BHW Plus Movies
Number analyzed (Participants) | 13 | 1
seconds
  Computerized Tower of London (cTOL) total time week 1 | 27.79 (5.79) | 26.78 (0)
  Computerized Tower of London (cTOL) total time week 11 | 25.21 (5.07) | 22.44 (0)
  Computerized Tower of London (cTOL) total time week 36: number analyzed (Participants) | 11 | 1
  Computerized Tower of London (cTOL) total time week 36 | 21.73 (3.08) | 26.78 (0)

2. Primary Outcome: Test of Grocery Shopping Skills
Description: Total time, week 1 and week 11 on a task of shopping in a local grocery store for 10 items as efficiently as possible, while selecting the correct size and cheapest unit cost. Total time with lower times=better performance.
Time Frame: week 1, 11
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | GMT Plus Attention | BHW Plus Movies
Number analyzed (Participants) | 13 | 1
minutes
  Test of grocery shopping skills week 1 | 24.34 (9.16) | 14.05 (0)
  Test of grocery shopping skills week 11 | 22.356 (9.07) | 13.12 (0)

3. Secondary Outcome: Attention Network Task
Description: Flanker task that dissociates attention into three components: alerting, orienting and executive control. Attention network effects were calculated using the following mean response time (RT) subtractions: alerting effect = no-cue RT minus center cue RT; orienting effect = invalid spatial cue RT minus valid spatial cue RT; executive control (conflict) effect = incongruent RT minus congruent RT. Mean response time for week 1, week 11 and week 36 on each component., lower=better performance.
Time Frame: week 1, 11, 36
Population: BHW participant 36 week Attention Network Task was not assessed.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | GMT Plus Attention | BHW Plus Movies
Number analyzed (Participants) | 14 | 1
milliseconds
  Attention Network Task Alerting, week 1 | 9.79 (30.04) | 38 (0)
  Attention Network Task Alerting week 11 | 39.39 (22.50) | 22 (0)
  Attention Network Task Alerting week 36: number analyzed (Participants) | 14 | 0
  Attention Network Task Alerting week 36 | 31.54 (15.88) |
  Attention Network Task Orienting week 1 | 57.61 (31.65) | 21 (0)
  Attention Network Task Orienting week 11 | 51.21 (31.65) | 15 (0)
  Attention Network Task Orienting week 36: number analyzed (Participants) | 14 | 0
  Attention Network Task Orienting week 36 | 46.21 (30.50) |
  Attention Network Task EC week 1 | 130.96 (64.88) | 145.5 (0)
  Attention Network Task EC week 11 | 80.68 (56.48) | 127 (0)
  Attention Network Task EC week 36: number analyzed (Participants) | 14 | 0
  Attention Network Task EC week 36 | 83.29 (29.22) |

4. Secondary Outcome: Community Reintegration of Service Members
Description: week 1, 11 and to week 36. The scale for each of the 46 items ranged from 1=extremely unsatisfied to 5=extremely satisfied. The total score is the mean of the responses of 46 items X 10. The range is 10 to 50 with higher numbers indicating better satisfaction with participation in the community.
Time Frame: week 1, 11, 36
Population: week 36 was not assessed for the BHW participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GMT Plus Attention | BHW Plus Movies
Number analyzed (Participants) | 13 | 1
score on a scale
  Community Reintegration of Service members Satisfaction week 1 | 23.23 (7.11) | 28.8 (0)
  Community Reintegration of Service members Satisfaction week 11 | 27.97 (7.02) | 29.29 (0)
  Community Reintegration of Service members Satisfaction week 36: number analyzed (Participants) | 13 | 0
  Community Reintegration of Service members Satisfaction week 36 | 27.59 (9.62) |

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | GMT Plus Attention | BHW Plus Movies
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/2
Other Adverse Events (participants affected / at risk) | 0/18 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT04044456/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT04044456/ICF_000.pdf